CLINICAL TRIAL: NCT04142411
Title: Combined Effect of Insulin and Sodium Hyaluronate Injection Guided by Ultrasound in Carpal Tunnel Syndrome
Acronym: PIT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Osama Aboshaera, Assistant Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AssiutUKAboshaera01
Record Dates: First submitted 2019-10-18; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Insulin; Hyaluronic Acid; Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Insulin and Sodium Hyaluronate Ultrasound guided injection (Experimental): Subjects will receive Ultrasound guided injection of 10 IU of crystalline insulin and 20 mg of Sodium Hyaluronate
  Interventions: Drug: Insulin; Drug: Sodium Hyaluronate; Device: Ultrasound
- Insulin Ultrasound guided injection (Active Comparator): Subjects will receive Ultrasound guided injection of 10 IU of crystalline insulin
  Interventions: Drug: Insulin; Device: Ultrasound
- Sodium Hyaluronate Ultrasound guided injection (Active Comparator): Subjects will receive Ultrasound guided injection of 20 mg of Sodium Hyaluronate
  Interventions: Drug: Sodium Hyaluronate; Device: Ultrasound

INTERVENTIONS:
Drug: Insulin — Ultrasound guided perineural injection therapy (PIT)
  Other Names: Crystalline Insulin
  Arms: Insulin Ultrasound guided injection; Insulin and Sodium Hyaluronate Ultrasound guided injection
Drug: Sodium Hyaluronate — Ultrasound guided perineural injection therapy (PIT)
  Other Names: Hyalgan
  Arms: Insulin and Sodium Hyaluronate Ultrasound guided injection; Sodium Hyaluronate Ultrasound guided injection
Device: Ultrasound — Philips Neuromuscular Ultrasound

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. The technique of perineural injection therapy (PIT) is now commonly used for peeling the nerve from surrounding soft tissue (called nerve hydrodissection), which may help to reduce neuro-inflammation, ischemic damage and allow impulse transmission.

The objective of this study is to evaluate the efficacy of ultrasound guided insulin plus Sodium Hyaluronate injection in reducing symptoms caused by carpal tunnel syndrome.

DETAILED DESCRIPTION:
In this randomized clinical trial, 90 patients with both a clinical and electromyographic diagnosis of mild to moderate carpal tunnel syndrome will be recruited from Assiut University Hospital (AUH). After obtaining written informed consent, patients will be randomized into three groups. Group A, patients will receive ultrasound-guided PIT with 10 IU of crystalline insulin; Group B, patients will receive ultrasound-guided PIT with 20 mg of Sodium Hyaluronate; Group C, patients will receive ultrasound-guided PIT with 10 IU of crystalline insulin and 20 mg of Sodium Hyaluronate. The primary outcome will be the Boston Carpal Tunnel Syndrome Questionnaire - Symptom Severity Scale at baseline, 1 month and 3 months post injection. All participants, investigator, outcomes assessor will be blinded (Triple blind)

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65
* Understanding written and spoken Arabic consent
* Diagnostic of carpal tunnel syndrome: Classic of probable based on the Katz Hand Diagram and mild to moderate based on the electrodiagnosis studies

Exclusion Criteria:

* Diseases known to cause carpal tunnel syndrome: Diabetes mellitus, hypothyroidism, connective tissue disease, rheumatic disease and moderate or severe chronic renal impairment
* Secondary diagnosis based on the ultrasound: arthrosynovial cyst, flexor tenosynovitis, ganglion
* Constant symptoms in medial nerve area
* Thenar eminence atrophy
* Cervical radiculopathy
* Brachial plexopathy
* Thoracic outlet syndrome
* Polyneuropathy
* Pregnancy
* Cognitive disorder
* Anticoagulant therapy
* Carpal tunnel injection in the last 6 months
* Ancient ipsilateral wrist fracture
* Ancient ipsilateral wrist surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire - Symptom Severity Scale | Baseline, 1 month, 3 months
  Boston carpal tunnel syndrome questionnaire - SSS is patient-based questionnaire for measurement of CTS severity which include11 questions to evaluate the symptom severity. Each question ranges from 1 to 5 with a higher score indicating a higher degree of disability.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire - Functional Status Scale | Baseline, 1 month, 3 months
  Boston carpal tunnel syndrome questionnaire - FSS is patient-based questionnaire for measurement of CTS functional disability which include 8 items to evaluate the functional status scale (FSS). Each item ranges from 1 to 5 with a higher score indicating a higher degree of disability.
Neuropathic pain Visual Analog Scale (VAS) | Baseline, 1 month, 3 months
  Digital pain severity or paresthesia/dysthesia was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.
U/S measured medial nerve mean CSA | Baseline, 1 month, 3 months
  Ultrasound measured medial nerve mean cross sectional area at the Pisiform bone level
U/S measured medial nerve CSA difference | Baseline, 1 month, 3 months
  Ultrasound measured medial nerve cross sectional area difference between pronator
U/S hyper-vascularization of medial nerve percentage | Baseline, 1 month, 3 months
  Percentage of Ultrasound hyper-vascularization of medial nerve in carpal tunnel
Sensory nerve conduction velocity of the median nerve | Baseline, 1 month, 3 months
  Antidromic sensory nerve conduction velocity of the median nerve

OTHER OUTCOMES:
Patient satisfaction (Likert scale) | 1month, 3 months
  Likert scale with the grade 1 means that the patient's satisfaction was 30%, grade 2, the patient's satisfaction was 30-50%, grade 3, the satisfaction was 50-80%, and grade 4 was 80%, Grades 3 and 4 were defined as "overall satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Khaled O Aboshaera, MD, Principal Investigator — Assistant Professor
Locations (1):
- Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith J, Wisniewski SJ, Finnoff JT, Payne JM. Sonographically guided carpal tunnel injections: the ulnar approach. J Ultrasound Med. 2008 Oct;27(10):1485-90. doi: 10.7863/jum.2008.27.10.1485. PMID 18809959
- [Background] Kamel SR, Sadek HA, Hamed A, Sayed OA, Mahmud MH, Mohamed FA, El Sagher GM, Aly LH. Ultrasound-guided insulin injection for carpal tunnel syndrome in type 2 diabetes mellitus patients. Clin Rheumatol. 2019 Oct;38(10):2933-2940. doi: 10.1007/s10067-019-04638-7. Epub 2019 Jun 17. PMID 31209710
- [Background] Apel PJ, Ma J, Callahan M, Northam CN, Alton TB, Sonntag WE, Li Z. Effect of locally delivered IGF-1 on nerve regeneration during aging: an experimental study in rats. Muscle Nerve. 2010 Mar;41(3):335-41. doi: 10.1002/mus.21485. PMID 19802878
- [Background] Ten Broek RPG, Stommel MWJ, Strik C, van Laarhoven CJHM, Keus F, van Goor H. Benefits and harms of adhesion barriers for abdominal surgery: a systematic review and meta-analysis. Lancet. 2014 Jan 4;383(9911):48-59. doi: 10.1016/S0140-6736(13)61687-6. Epub 2013 Sep 27. PMID 24075279